CLINICAL TRIAL: NCT04772079
Title: A Multicenter, Randomized, Double-Blind Placebo-Controlled Phase 3 Study to Evaluate the Pharmacokinetics, Efficacy and Safety of Deucravacitinib (BMS-986165) in Pediatric Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Evaluate the Drug Levels, Efficacy and Safety of Deucravacitinib in Pediatric Participants With Moderate to Severe Plaque Psoriasis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM011-126; 2019-004879-39 (EudraCT Number)
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Plaque Psoriasis
Keywords: Adolescent Psoriasis; BMS-986165; Clinical trial; Deucravacitinib; Pediatric; Pediatric Psoriasis; Plaque Psoriasis; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Active treatment deucravacitinib standard dose (Experimental)
  Interventions: Drug: Deucravacitinib
- Active treatment deucravacitinib half-standard dose (Experimental)
  Interventions: Drug: Deucravacitinib
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo matching deucravacitinib

INTERVENTIONS:
Drug: Deucravacitinib — Specified dose on specified days
  Arms: Active treatment deucravacitinib half-standard dose; Active treatment deucravacitinib standard dose
Other: Placebo matching deucravacitinib — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this pediatric study is to evaluate the drug levels, efficacy and safety of Deucravacitinib in pediatric participants aged 4 to <18 years with moderate to severe plaque psoriasis. This study includes two cohorts; Cohort 1 (age 12 to <18 years) and Cohort 2 (age 4 to <12 years), with two parts; for each cohort. Part A will evaluate the drug levels of BMS-986165 to enable selection of 2 dose levels to be studied in Part B. Part B will assess the efficacy and safety of two dose levels in pediatric participants with moderate to severe plaque psoriasis. The 5-year long-term extension (LTE) period will observe the long-term safety and tolerability of deucravacitinib in pediatric participants with psoriasis who have completed Parts A or B of the study.

ELIGIBILITY:
Inclusion Criteria

* Males and females aged 12 to <18 years for Cohort 1. Males and females aged 4 to <12 years for Cohort 2.
* Plaque psoriasis for at least 6 months.
* Moderate to severe disease.
* Candidate for phototherapy or systemic therapy.
* Must have completed the Week 52 treatment period in Part A or B for long-term extension (LTE) period.

Exclusion Criteria

* Participants weighing ≤ 30.0 kg at screening for Cohort 1 (age 12 to < 18 years), Part A and Part B. Participants weighing ≤ 18.0 kg at screening for Cohort 2 (age 4 to < 12 years), Part A and Part B.
* Other forms of psoriasis.
* History of recent infection.
* Prior exposure to deucravacitinib (BMS-986165) or active comparator.
* Evidence of active TB for LTE period.
* Other protocol-defined inclusion/exclusion criteria apply.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 153 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2033-09-08 (Estimated)

PRIMARY OUTCOMES:
Geometric mean observed average concentration at steady state (Cavg.ss) for deucravacitinib at Week 2 | Week 2
  Part A
Maximum observed plasma concentration at steady state (Cmax.ss) for deucravacitinib at Week 2 | Week 2
  Part A
Trough observed plasma concentration (Ctrough) for deucravacitinib at Week 2 | Week 2
  Part A
Proportion of subjects with at least 75% improvement in Psoriasis Area and Severity Index (PASI 75) at Week 16 | Week 16
  Part B
Proportion of subjects with an static Physician's Global Assessment (sPGA) score of 0 (clear) or 1 (almost clear) with at least a 2-point reduction from baseline at Week 16 | Week 16
  Part B
Incidence of Adverse Events (AEs) | Up to 316 weeks
  Long-term extension (LTE) Period
Incidence of serious adverse events (SAEs) | Up to 316 weeks
  LTE Period
Monitoring of growth: Body weight | Up to 316 weeks
  LTE Period
Monitoring of growth: Height | Up to 316 weeks
  LTE Period
Monitoring of growth: Tanner staging (sexual maturation) | Up to 316 weeks
  LTE Period

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 424 days
  Part A and Part B
Incidence of serious adverse events (SAEs) | Up to 466 days
  Part A and Part B
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Up to 466 days
  Part A and Part B
Incidence of clinically significant changes in clinical laboratory results: Chemistry panel tests | Up to 466 days
  Part A and Part B
Incidence of clinically significant changes in clinical laboratory results: Urinalysis tests | Up to 466 days
  Part A and Part B
Incidence of clinically significant changes in clinical laboratory results: Hemoglobin A1C tests | Up to 410 days
  Part A and Part B
Incidence of clinically significant changes in clinical laboratory results: Infectious serologies tests | Up to 42 days
  Part A and Part B
Incidence of clinically significant changes in clinical laboratory results: Tuberculosis (TB) tests | Up to 42 days
  Part A and Part B
Incidence of clinically significant changes in clinical laboratory results: Lipid panel tests | Up to 368 days
  Part A and Part B
Incidence of clinically significant changes in clinical laboratory results: Serum immunoglobulin level tests | Up to 368 days
  Part A and Part B
Incidence of clinically significant changes in clinical laboratory results: Fasting plasma glucose tests | Up to 368 days
  Part A and Part B
Incidence of clinically significant changes in clinical laboratory results: Pregnancy test for women of childbearing potential only | Up to 466 days
  Part A and Part B
Incidence of clinically significant changes in lymphocyte subsets and function | Up to 466 days
  Part A and Part B
Incidence of clinically significant changes in cytokine levels | Up to 466 days
  Part A and Part B
Incidence of clinically significant changes in physical examination findings | Up to 466 days
  Part A and Part B
Incidence of clinically significant changes in vital signs: Body temperature | Up to 466 days
  Part A and Part B
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 466 days
  Part A and Part B
Incidence of clinically significant changes in vital signs: Systolic and diastolic blood pressure | Up to 466 days
  Part A and Part B
Incidence of clinically significant changes in vital signs: Heart rate | Up to 466 days
  Part A and Part B
Monitoring of growth: Body weight | Up to 466 days
  Part A and Part B
Monitoring of growth: Height | Up to 466 days
  Part A and Part B
Monitoring of growth: Tanner staging (sexual maturation) | Up to 466 days
  Part A and Part B
Proportion of subjects with at least 75% improvement in PASI (PASI 75) at Week 16 for the comparison of the half-standard dose of deucravacitinib vs placebo | Week 16
  Part B
Proportion of subjects with an sPGA score of 0 (clear) or 1 (almost clear) with at least a 2-point reduction from baseline at Week 16 for the comparison of the half-standard dose of deucravacitinib vs placebo | Week 16
  Part B
Proportion of subjects with at least 90% improvement in PASI (PASI 90) at Week 16 for the comparison of deucravacitinib vs placebo | Week 16
  Part B
Change from baseline in PASI at Week 16 for comparison of deucravacitinib vs placebo | Week 16
  Part B
Change from baseline in BSA involvement at Week 16 for comparison of deucravacitinib vs placebo | Week 16
  Part B
Change from baseline in CDLQI score at Week 16 for comparison of deucravacitinib vs placebo | Week 16
  Part B
Change from baseline in subject reported visual analog scale (VAS) for subject's assessment of joint pain at Week 16 (only for subjects with confirmed JPsA prior to baseline) for comparison of deucravacitinib vs placebo | Week 16
  Part B
Change from baseline in VAS for subject's Global Assessment of Joint Disease; at Week 16 (only for subjects with confirmed JPsA prior to baseline) for comparison of deucravacitinib vs placebo | Week 16
  Part B
Proportion of subjects achieving American College of Rheumatology Pediatric 30 (ACR Pedi 30) response at Week 16 for subjects with confirmed JPsA prior to baseline | Week 16
  Part B
  ACR Pedi 30 response is defined as subjects with at least 30% improvement from baseline in 3 of any 6 variables in the core set, while no more than one of the remaining variables can worsen by > 30% for comparison of deucravacitinib vs placebo
Proportion of subjects using topical corticosteroid at Week 16 for comparison of deucravacitinib vs placebo | Week 16
  Part B
Proportion of subjects with protective titers of antibodies to measles, tetanus and pertussis at Week 16 | Week 16
  Part B
Geometric mean observed average concentration at steady state (Cavg.ss) for deucravacitinib at Week 16 | Week 16
  Part B
Maximum observed plasma concentration at steady state (Cmax.ss) for deucravacitinib at Week 16 | Week 16
  Part B
Trough observed plasma concentration (Ctrough) for deucravacitinib at Week 16 | Week 16
  Part B
Proportion of participants with 75% improvement in PASI (PASI 75) over time | Up to 316 weeks
  LTE Period
Proportion of participants with an sPGA score of 0 (clear) or 1 (almost clear) with at least a 2-point reduction from baseline over time | Up to 316 weeks
  LTE Period

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (63):
- Argentina (6):
  - Instituto de Neumonologia Y Dermatologia, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Psoriahue, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - CONEXA Investigacion Clinica S.A., Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - Hospital Italiano de Buenos Aires, CABA
  - Consultora Integral de Salud, Córdoba
- Australia (6):
  - The Skin Hospital, Darlinghurst, New South Wales
  - Local Institution - 0002, Westmead, New South Wales
  - Queensland Children's Hospital, Brisbane, Queensland
  - Veracity Clinical Research, Woolloongabba, Queensland
  - Monash Health, Clayton, Victoria
  - Local Institution - 0001, Melbourne, Victoria
- Brazil (5):
  - Centro de Pesquisas da Clínica IBIS, Salvador, Estado de Bahia
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo (USP) - HCFMRP, Ribeirão Preto, São Paulo
  - Local Institution - 0083, Rio de Janeiro
  - Local Institution - 0067, São Paulo
- Canada (5):
  - Local Institution - 0010, Calgary, Alberta
  - Alberta Dermasurgery Centre, Edmonton, Alberta
  - Local Institution - 0039, Hamilton, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
- France (4):
  - Centre Hospitalier de Calais, Calais
  - Centre Hospitalier Universitaire Dijon Bourgogne - Hôpital François Mitterrand-dermatology, Dijon
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet, Nice
  - Local Institution - 0021, Paris
- Germany (5):
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsmedizin Johannes Gutenberg Universität Mainz, Mainz, Rhineland-Palatinate
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden, Saxony
  - Charité Universitaetsmedizin Berlin - Campus Mitte, Berlin
  - Kath. Kinderkrankenhaus Wilhelmstift, Hamburg
- Japan (7):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Fukuoka University Hospital, Fukuoka, Jonan-Ku, Fukuoka
  - Local Institution - 0040, Isehara, Kanagawa
  - Mie University Hospital, Tsu, Mie-ken
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Nippon Life Hospital, Osaka
- Mexico (4):
  - Crea de Guadalajara, Guadalajara, Jalisco
  - Grupo Clínico CATEI S.C., Guadalajara, Jalisco
  - RM Pharma Specialists, Mexico City, Mexico City
  - Arké SMO S.A de C.V, Veracruz
- Poland (4):
  - Local Institution - 0011, Krakow
  - Dermoklinika Centrum Medyczne S.C. M. Kierstan, J. Narbutt, A. Lesiak, Lodz
  - Państwowy Instytut Medyczny MSWiA-Klinika Dermatologii, Warsaw
  - WroMedica, Wroclaw
- Romania (7):
  - Local Institution - 0080, Bucharest, București
  - Local Institution - 0081, Bucharest, București
  - Local Institution - 0088, Bucharest, București
  - CCBR Clinical Research, Bucharest, București
  - Lotus-Med Tunari, Bucharest
  - Spitalul clinic de urgenta pentru copii Sf. Maria, Iași
  - Spitalul Clinic Judetean Mures, Târgu Mureş
- South Korea (3):
  - Local Institution - 0048, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0047, Seoul, Seoul-teukbyeolsi [Seoul]
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
- Spain (6):
  - Hospital General Universitario de Alicante-Dermatology, Alicante
  - OSI Ezkerraldea-Enkarterri-Cruces - Hospital Universitario Cruces-Dermatology, Barakaldo
  - Hospital Sant Joan de Déu-URC Dermatology, Esplugues de Llobregat
  - Hospital Universitario de Gran Canaria Doctor Negrín-Dermatología, Las Palmas de GC
  - Hospital Universitario 12 de Octubre-DERMATOLOGY, Madrid
  - Hospital Universitario La Paz-UCICEC/DERMA, Madrid
- Mounts Bay Medical, Connor Downs, United Kingdom

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04772079.html